CLINICAL TRIAL: NCT03419247
Title: Comprehensive Molecular Profiling of Advanced Biliary Tract Cancers (BTC) for Better Treatment Selection: A Prospective Study (COMPASS B)
Brief Title: Molecular Profiling of Advanced Biliary Tract Cancers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not activated
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COMPASS-B
Record Dates: First submitted 2017-12-07; First posted 2018-02-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor tissue and blood sample collection (Experimental)
  Interventions: Procedure: Fresh tumor tissue biopsy; Procedure: Blood draw; Procedure: Archival tumor tissue collection

INTERVENTIONS:
Procedure: Fresh tumor tissue biopsy — A type of surgical procedure that will use a thin needle to remove a sample of tumor tissue.
Procedure: Blood draw — Blood will be taken by a needle from a vein.
Procedure: Archival tumor tissue collection — A sample of tumor tissue that was taken by biopsy or surgery before agreeing to take part in this study will be collected.

SUMMARY:
This is a study where fresh tumor tissue and blood samples will be collected from patients with advanced biliary tract cancer who will be undergoing 1st line therapy with gemcitabine or fluorouracil (5-FU) regimens to see how useful it is to look for changes and characteristics in genes (molecules that contain instructions for the development and functioning of the cells) and the genes within the tumour to find characteristics that may be useful in choosing treatments for patients in the future.

DETAILED DESCRIPTION:
Changes (mutations) in genes have been shown to be an important characteristic in cancers. Looking at differences in genes in patients with unresectable or metastatic biliary tract cancer and comparing this information with response to their initial chemotherapy treatment may help to learn which treatments may be better for certain patients after initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological or radiological diagnosis of inoperable or metastatic biliary tract cancer (BTC).
* Patient must have a tumor lesion that is amenable to a core needle biopsy as judged by a staff radiologist.
* Patients must have a measurable lesion by RECIST 1.1 in addition to the lesion that is going to be biopsied.
* Patients must be fit enough to safely undergo a tumor biopsy as judged by the investigator.
* Eastern Cooperative Group (ECOG) performance status ≤ 1 (Karnofsky ≥60%).
* Life expectancy of greater than 90 days, as judged by the investigator.
* Within 14 days of the proposed biopsy date, patients must have normal organ and marrow function.
* Patients must undergo systemic treatment with gemcitabine or 5-FU based regimens as first line standard systemic palliative treatment with or without other investigational agents within a clinical trial.
* Ability to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patients with one or more contraindications to tumor biopsy.
* Patients who have had prior systemic treatment (chemotherapy or any other anti-cancer agent) in the advanced setting.
* Patients who are currently on anti-cancer treatment including chemotherapy.
* Patients with known brain metastases are excluded from participation in this clinical study.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-01-02 (Estimated); Study Completion 2023-01-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with gene testing data available at 8 weeks from baseline tumor biopsy. | 8 Weeks

SECONDARY OUTCOMES:
Disease control rate | 4 years
Progression-free survival rate | 4 years
Overall survival rate | 4 years
Genomic predictors of response to chemotherapy identified | 4 years
Germline mutations of hereditary risk factors | 4 years
Potential predictive biomarkers of response to treatment such as BRCA, PALB2 and ATM mutations. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Knox, M.D., Principal Investigator — Princess Margaret Cancer Centre

IPD SHARING:
Plan to Share IPD: No